CLINICAL TRIAL: NCT07361419
Title: Metabolic Response to Supine Physiotherapy in Mechanically Ventilated Critically Ill Patients Assessed by Indirect Calorimetry
Brief Title: Metabolic Response to Supine Physiotherapy in Mechanically Ventilated ICU Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Universidad de Extremadura (Other)
Responsible Party: Principal Investigator, Carlos Fernández-Morales, Clinical Professor, Universidad de Extremadura
Other Study IDs: 12
Record Dates: First submitted 2026-01-14; First posted 2026-01-23 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Critical Illness; Mechanical Ventilation; Intensive Care Unit-Acquired Weakness; Physical Rehabilitation in the Intensive Care Unit
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Passive Supine Physiotherapy: Adult critically ill patients receiving invasive mechanical ventilation who undergo standardized passive supine physiotherapy as part of usual ICU care. During the physiotherapy session, oxygen consumption is continuously measured using indirect calorimetry integrated into the ventilator, including baseline rest, intervention, and recovery periods.
  Interventions: Procedure: Supine Physiotherapy Session
- Active-Assisted Supine Physiotherapy: Adult critically ill patients receiving invasive mechanical ventilation who undergo active-assisted supine physiotherapy as part of usual intensive care unit care. Physiotherapy consists of active-assisted limb mobilization, in which the patient voluntarily initiates the movement and the physiotherapist provides assistance as needed to complete the range of motion. This intervention is applied in patients who are awake or lightly sedated and able to cooperate.
  Interventions: Procedure: Supine Physiotherapy Session

INTERVENTIONS:
Procedure: Supine Physiotherapy Session — Adult critically ill patients receiving invasive mechanical ventilation who undergo passive supine physiotherapy as part of usual intensive care unit care. Physiotherapy consists exclusively of passive limb mobilization performed by a physiotherapist, with no voluntary muscle activation by the patient, and is applied in deeply sedated patients.

SUMMARY:
Critically ill patients who require mechanical ventilation frequently experience rapid loss of muscle mass and physical function during their stay in the intensive care unit (ICU). As part of standard care, physiotherapy and limb mobilization exercises are commonly provided, even in patients who are sedated and confined to bed in a supine position. However, the actual physiological and metabolic intensity of these routine physiotherapy interventions is poorly understood, and current prescriptions are largely based on clinical judgment rather than objective measures of patient effort or tolerance.

Oxygen consumption (VO₂) is a direct indicator of metabolic demand and physiological workload. In mechanically ventilated patients, indirect calorimetry integrated into the ventilator allows continuous measurement of VO₂ and carbon dioxide production without adding invasive procedures. While indirect calorimetry is routinely used to individualize nutritional support in the ICU, its potential role in quantifying the metabolic cost of physiotherapy interventions has been scarcely explored.

The aim of this prospective observational study is to quantify the acute metabolic response to a standardized session of supine physiotherapy in adult critically ill patients receiving invasive mechanical ventilation. During routine physiotherapy sessions performed as part of usual care, oxygen consumption will be continuously measured using indirect calorimetry integrated into the ventilator circuit. Each session will include a baseline resting period, the physiotherapy intervention itself, and a post-intervention recovery period, allowing patients to act as their own controls.

Physiotherapy sessions will consist of passive limb mobilization in deeply sedated patients and passive or active-assisted mobilization in patients who are awake or lightly sedated and able to cooperate. The primary outcome will be the change in oxygen consumption during physiotherapy compared with baseline rest. Secondary analyses will describe the total metabolic load of the session, peak oxygen consumption, and the time required for oxygen consumption to return toward baseline levels after the intervention. Basic cardiorespiratory variables, such as heart rate, blood pressure, oxygen saturation, and ventilatory parameters, will also be recorded to assess physiological stability and tolerance.

By objectively characterizing the metabolic cost of common supine physiotherapy interventions, this study aims to improve understanding of the physiological demands imposed on mechanically ventilated ICU patients. The results may help inform safer and more individualized physiotherapy prescriptions in critical care, supporting a more objective approach to dosing rehabilitation based on patients' real metabolic responses rather than solely on activity type or sedation level.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.

Admission to the intensive care unit.

Invasive mechanical ventilation via endotracheal tube or tracheostomy.

Ability to remain in the supine position during the measurement period.

Clinical indication for supine physiotherapy as part of usual ICU care.

Richmond Agitation-Sedation Scale (RASS) score between -5 and 0 at the time of the session.

Hemodynamic stability, defined as mean arterial pressure ≥65 mmHg with or without vasopressor support and no initiation or increase >20% in vasopressor dose within the previous 60 minutes.

Respiratory stability, defined as no changes in ventilator settings within the previous 30 minutes and oxygen saturation ≥90% with FiO₂ ≤0.60 and PEEP ≤12 cmH₂O.

Technical conditions allowing valid indirect calorimetry measurement (absence of significant air leaks and no planned circuit disconnections).

Exclusion Criteria:

* Use of extracorporeal membrane oxygenation (ECMO) or other extracorporeal gas exchange systems.

Continuous renal replacement therapy during the measurement period when it may interfere with metabolic measurements.

Significant air leaks in the airway or ventilator circuit that invalidate indirect calorimetry measurements.

Planned procedures or interventions during the measurement period that could interfere with gas exchange (e.g., bronchoscopy, recruitment maneuvers, ventilator setting changes).

Severe respiratory instability requiring FiO₂ >0.60 or PEEP >12 cmH₂O.

Ongoing neuromuscular blockade infusion.

Clinical contraindications to limb mobilization (e.g., unstable fractures, active bleeding, uncontrolled intracranial hypertension).

Agitation or risk of unplanned device removal (RASS >0).

Refusal of participation by the patient or legally authorized representative, when applicable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult critically ill patients admitted to the intensive care unit who require invasive mechanical ventilation and receive routine supine physiotherapy as part of standard care. The study population includes both deeply sedated patients undergoing passive mobilization and awake or lightly sedated patients able to perform active-assisted mobilization, allowing characterization of metabolic responses across different levels of consciousness and participation.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in Oxygen Consumption (ΔVO₂) During Supine Physiotherapy | During a single physiotherapy session (baseline rest and intervention periods).
  Oxygen consumption (VO₂) will be continuously measured using indirect calorimetry integrated into the mechanical ventilator during a standardized supine physiotherapy session performed as part of usual ICU care. The primary outcome is the change in VO₂ (ΔVO₂), defined as the difference between mean VO₂ during the physiotherapy intervention and mean VO₂ during a preceding baseline resting period, within the same session. Each participant serves as their own control.

SECONDARY OUTCOMES:
Total Metabolic Load of the Physiotherapy Session (VO₂ Area Under the Curve Above Baseline) | During a single physiotherapy session (baseline, intervention, and recovery periods)
  Oxygen consumption (VO₂) will be continuously measured by indirect calorimetry during baseline rest, the physiotherapy intervention, and the recovery period. Total metabolic load will be expressed as the area under the VO₂-time curve above baseline (AUC above baseline), integrating the excess VO₂ over time attributable to the session.
Peak Oxygen Consumption During Supine Physiotherapy | During the physiotherapy intervention period of a single session
  Peak VO₂ will be defined as the highest VO₂ value observed during the physiotherapy intervention period, measured continuously via indirect calorimetry. The outcome will be reported as the absolute peak VO₂ and may be expressed relative to baseline.
Relative Change in Oxygen Consumption During Supine Physiotherapy (%ΔVO₂) | During a single physiotherapy session (baseline rest and intervention periods).
  The relative change in oxygen consumption will be calculated as the percentage difference between mean VO₂ during the physiotherapy intervention and mean VO₂ during baseline rest within the same session.
Time to Recovery of Oxygen Consumption Toward Baseline After Physiotherapy | Immediately after the physiotherapy intervention, up to the end of the recovery monitoring period within a single session.
  Recovery time will be defined as the time required after the end of the physiotherapy intervention for VO₂ to return to within ±10% of the baseline mean value and remain within that range for a sustained period (as per protocol). If VO₂ does not return to this range within the maximum monitoring window, recovery will be recorded as not achieved within the session.
Cardiorespiratory Stability During Supine Physiotherapy | During a single physiotherapy session (baseline, intervention, and recovery periods).
  Physiological stability during the session will be assessed by changes from baseline in heart rate, blood pressure (including mean arterial pressure), peripheral oxygen saturation (SpO₂), and ventilatory parameters recorded during baseline rest, intervention, and recovery. Clinically relevant events leading to interruption of the session (e.g., desaturation, hypotension, arrhythmia) will be documented.
Carbon Dioxide Production (VCO₂) and Respiratory Exchange Ratio (RER) During Supine Physiotherapy | During a single physiotherapy session (baseline, intervention, and recovery periods).
  Carbon dioxide production (VCO₂) will be continuously measured by indirect calorimetry during baseline rest, intervention, and recovery. Respiratory exchange ratio (RER) will be calculated as VCO₂/VO₂ for the same periods to describe metabolic response patterns.
Energy Expenditure During Supine Physiotherapy | During a single physiotherapy session (baseline, intervention, and recovery periods).
  Energy expenditure will be estimated from VO₂ and VCO₂ as provided by the indirect calorimetry system. Values will be summarized for baseline rest, the physiotherapy intervention, and the recovery period within the same session.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Badajoz, Badajoz, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: No